CLINICAL TRIAL: NCT00873782
Title: Safety and Feasibility of Transvenous Limb Perfusion With Normal Saline in Human Muscular Dystrophy
Brief Title: Safety Study of Transvenous Limb Perfusion in Human Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of North Carolina (Other)
Responsible Party: Principal Investigator, William Powers, Professor of Neurology, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U54AR056953 (NIH); U54AR056953 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-01

CONDITIONS: Muscular Dystrophies; Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Limb-Girdle Muscular Dystrophy
Keywords: Limb Perfusion; Gene Therapy
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Dystrophies, Limb-Girdle | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will undergo retrograde high pressure transvenous limb perfusion with normal saline.
  Interventions: Other: Retrograde high pressure transvenous perfusion with normal saline

INTERVENTIONS:
Other: Retrograde high pressure transvenous perfusion with normal saline — Dose escalation of saline volume, infusion rate, and tourniquet pressure, as determined in a stepwise manner and by careful monitoring

SUMMARY:
Muscular dystrophies are inherited disorders in which the skeletal and heart muscles become progressively weaker, sometimes leading to permanent disability. Current treatments aim to control symptoms as much as possible, but there is no cure. Gene therapy, in which defective genes causing the disorder are corrected, is a potential treatment option and is in the process of being developed for muscular dystrophies. This study will determine the safety and feasibility of a particular delivery method for gene therapy that could be used in the future to treat people with muscular dystrophies. Only normal saline, and no active treatment, will be used in this study.

DETAILED DESCRIPTION:
There are many types of muscular dystrophies, all of which are progressive, degenerative genetic disorders. One type is Becker's muscular dystrophy, which involves slowly worsening muscle weakness of the legs and pelvis and which can lead to cardiomyopathy, deformities, respiratory failure, and permanent disability. Limb-girdle muscular dystrophy, another type, is also characterized by progressive muscle weakness, first affecting the muscles around the shoulder girdle and hips and possibly affecting other muscles as the disorder progresses. Complications of limb-girdle muscular dystrophy can include abnormal heart rhythms, joint contractures, difficulties with activities of daily living, significant loss of mobility, and permanent disability. There is no cure for muscular dystrophies. Current treatments, such as steroids, mobility aids, physical therapy, and respiratory care, can decrease some of the complications, but there is a clear need for a curative therapy.

The genetic basis of muscular dystrophies is well understood, which makes gene therapy a potential treatment option in the future. A key step in developing gene therapy involves first ensuring safe delivery of genetic material into a single limb of a patient before using active treatment in the patient's entire body. High-pressure, high-volume transvenous limb perfusion, in which fluid is forced under high pressure into arm and leg muscles through the veins, has shown the greatest potential as a delivery method. The purpose of this study is to determine the safety and feasibility of this method with normal saline in people who have Becker's muscular dystrophy or limb-girdle muscular dystrophy.

Participation in this study will last up to 4 weeks. At an initial baseline visit, participants will undergo water emersion measurements of their arm and leg, nerve testing, and muscle strength testing. About 1 to 2 weeks later, participants will enter the pediatric intensive care unit for up to 36 hours. During the inpatient stay, participants will undergo the high-pressure, high-volume transvenous limb perfusion procedure with normal saline in one of their arms or legs. Throughout the hospital stay, breathing, heart rate, and blood pressure will be monitored. Medication will be available to control any discomfort or pain experienced by participants. Each subsequent participant will receive more fluid pumped at a higher pressure and with a tighter tourniquet than the previous participant, as long as no problems or adverse effects are detected. Some of the participants will undergo an MRI immediately after the perfusion procedure. About 1 to 2 weeks after the inpatient stay, participants will attend a follow-up visit that will include repeat nerve and muscle strength testing, a blood draw, photos of limbs, and an ultrasound of the leg blood vessels if the participant's leg was used during the perfusion procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Duchenne or Becker muscular dystrophy, as defined by progressive weakness with onset before the age of 21, X-linked inheritance, and reduced dystrophin (less than 3%) on muscle biopsy OR mutation in the dystrophin gene
* Diagnosis of limb girdle muscular dystrophy, as defined by progressive weakness with onset before the age of 21, normal dystrophin on muscle biopsy OR proven mutation associated with one of the types of limb girdle dystrophy
* Older than 21 years of age and preferably younger 30 years of age
* Able to stand, independently or with assistance
* Able to communicate with pertinent staff
* Able to understand and willingly comply with the requirements of the study

Exclusion Criteria:

* Confirmed diagnosis of any other muscle disease
* Previous compartment syndrome requiring surgical decompression
* Previous venous or arterial thrombosis other than superficial venous thrombosis associated with intravenous catheter
* Coagulopathy, including known diagnosis of bleeding diathesis, history of excessive bleeding on multiple occasions, or taking anticoagulant or platelet inhibitory medications
* Systemic arterial or venous disease (e.g., Raynaud's, aortic coarctation or aneurysm)
* Previous injury to selected limb with residual effect other than superficial scarring
* Previous vascular surgery to selected limb
* Previous compressive neuropathy (e.g., carpal tunnel syndrome in arm, peroneal palsy in leg)
* Complex regional pain syndrome or other neurological cause of limb pain
* Previous clinical diagnosis of congestive heart failure
* Previous echocardiography showing ejection fraction less than 40% or ventricular dilation
* Previous chest x-ray showing enlarged cardiac silhouette or pulmonary edema
* History of rhabdomyolysis with worsening renal function
* Creatinine greater than 1.7 mg/dL
* Resting hypoxemia with SaO2 less than 90% on room air
* Other significant heart, lung, or kidney disease that would compromise the body's capacity to handle a fluid load
* Previous forced vital capacity less than 75% of age and height adjusted norm, in the absence of acute reversible pulmonary disease
* Sickle cell disease (sickle cell anemia [SS] or sickle hemoglobin C disease [SC])
* Pregnant
* Non-English speaker

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Powers, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Pressure Transvenous Limb Perfusion: Participants will undergo retrograde high pressure transvenous limb perfusion of an arm or a leg with normal saline through an 18g or 20g peripheral catheter with a tourniquet on the upper part of the limb: The volume of saline as % of perfused limb volume was escalated beginning at 5%. Safety was determined by Doppler ultrasound to assess venous and arterial damage electrodiagnostic neurographic testing quantitative muscle testing strength assessments, the Action Research Arm Test (ARAT), basic metabolic panel (Na+, K+, Cl-, CO2, BUN, and creatinine), serum creatine kinase [CK], plasma and urine myoglobin. Some subjects underwent MRI to assess whether saline went subcutaneously or intramuscularly.
Period: Overall Study
Arm/Group | High Pressure Transvenous Limb Perfusion
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High Pressure Transvenous Limb Perfusion
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Muscle, Nerve, or Vascular Damage
Description: Number of Participants with all of the following three:
  1. Unchanged Doppler ultrasound to assess venous and arterial damage pre-and post perfusion based on report
  2. Without clinically significant changes in electrodiagnostic testing using standard neurographic techniques pre-and post perfusion:>1 mSec change in baseline distal motor latency; <75% baseline compound muscle action potential amplitude, <75% baseline conduction velocity, sensory nerve action potential
  3. Without clinically significant changes in Quantitative muscle testing (QMT) strength assessments pre-and post perfusion:< 85% baseline
Time Frame: Measured within 2 weeks after limb perfusion procedure
Measure: Number; unit: participants
Arm/Group | High Pressure Transvenous Limb Perfusion
Number analyzed (Participants) | 16
participants | 16

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | High Pressure Transvenous Limb Perfusion
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 12/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Pressure Transvenous Limb Perfusion (N=16)
Ankle pain (Musculoskeletal and connective tissue disorders) | 2
Elevated Muscle Compartment pressures (Musculoskeletal and connective tissue disorders) | 10
Reduced Compound Muscle Action Potentials (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No